CLINICAL TRIAL: NCT05837975
Title: Effect of the Exoskeleton for Assisting Ambulatory Activities in People With Subacute Stroke : a Randomized, Cross-over Trial
Brief Title: Effect of the Exoskeleton for Assisting Ambulatory Activities in People With Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202319
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Exoskeleton
Keywords: Subacute; Motor function; Robot; Walking assistance; Home mobility aid
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FREE Walk Exoskeleton vs Traditional Rehabilitation for Stroke Patients (Experimental): Participants in this arm will receive one month of traditional rehabilitation followed by one month of using the exoskeleton at home.
  Interventions: Device: FREE Walk Exoskeleton; Other: Traditional Rehabilitation
- Traditional Rehabilitation vs FREE Walk Exoskeleton for Stroke Patients (Experimental): Arm Description: Participants in this arm will receive one month of using the exoskeleton at home followed by one month of traditional rehabilitation.
  Interventions: Device: FREE Walk Exoskeleton; Other: Traditional Rehabilitation

INTERVENTIONS:
Device: FREE Walk Exoskeleton — Using a robotic exoskeleton to help with lower limb activities that are difficult due to neurological diseases. Used at home for individual patient training.
Other: Traditional Rehabilitation — Traditional rehabilitation refers to the use of conventional therapeutic methods.

SUMMARY:
Background: Although rehabilitation activities, including physical therapy, are known to be beneficial for stroke patients, many patients still have poor walking function, especially after the acute phase of three months, where the recovery of lower limb walking ability through traditional rehabilitation therapy gradually decreases, requiring alternative approaches. Exoskeleton robots appear to provide benefits for stroke patients by providing exercise guidance, thus improving their independent gait endurance and stair climbing ability. For stroke patients who cannot continue to improve through general rehabilitation and have ongoing mobility difficulties, exoskeletons may be a potential solution. However, previous literature on the use of exoskeletons to assist gait training has had mixed results, with one major reason being that the frequency of use is too low or the duration of use is too short, due to the high cost and inconvenience of travel to medical institutions. Therefore, it is necessary to find ways to enable patients to use them frequently and for a long period.

Method: investigators designed a non-blinded, randomized crossover trial to observe the potential benefits of using the device at home for one month. Patients were randomly divided into two groups, one receiving traditional rehabilitation first and the other using the exoskeleton first. There were four time points for testing: before, after the first stage of treatment, after the second stage of treatment, and one month after completing the second stage, to observe the sustained effects.

The testing involved executing a 6-minute walk test, timed up and go test, and a 10-step stair test (up and down) both with and without the device. An electronic software app was used to record daily usage time to determine the quantity and degree of home use.

Analysis: Repeated measures ANOVA models were used to analyze the effects and correlations of the experiment. The effects of the duration/frequency of use on dosage were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with first-time stroke, with onset time within 1 month to 2 years from the time of recruitment, and all participants must sign an informed consent form.
2. Patients must have independent walking ability, with or without cane.
3. Lower limb muscle tone Modified Ashworth Scale <3.
4. Able to perform a 25-meter walking test and a 10-step stair test without assistance from others.
5. Cognitive function Mini-Mental State Examination > 23 points.

Exclusion Criteria:

1. Combined with other central nervous system problems, such as brain tumors or spinal cord injuries.
2. Clearly, lower limb joint diseases that cannot achieve complete hip, knee, and ankle joint activity are not excluded, but mild joint activity limitations caused by stroke are not excluded.
3. Skin diseases that are not suitable for contact with exoskeleton devices.
4. Unable to cooperate with the two-month research plan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
final distance walked by the 6-minute walk test | before, after the first stage of treatment, after the second stage of treatment, and one month after completing the second stage, to observe the sustained effects.
  Unit in meters, used to evaluate gait function and endurance. Participants walk along a 30-meter walkway, turning back within 6 minutes and recording the total distance covered at the end. Patients are allowed to rest during the test but not run. A higher score (walking distance) indicates better gait and endurance.This range overlaps with data reported in other populations.
Time difference of Timed up and go' test (TUG) | before, after the first stage of treatment, after the second stage of treatment, and one month after completing the second stage, to observe the sustained effects.
  The TUG test (time measured in seconds) is a common clinical test for mobility function, using the 3-meter TUG test and following the procedure of Podsiadlo and Richardson's standards. The method involves asking the patient to sit on a straight-backed chair, then stand up, walk three meters forward at their usual pace, turn around, and return to sit on the chair. The total time is recorded with a stopwatch. The test is repeated five times. For this test, a lower score (time to complete) means better overall mobility.
Time difference of 10-step stair test | before, after the first stage of treatment, after the second stage of treatment, and one month after completing the second stage, to observe the sustained effects.
  Timed Stair Test(TST) is a timed test measured in seconds, where the participant ascends and descends 10 steps of a staircase. The time taken to ascend(TSTup) and descend(TSTdn) is measured separately using a stopwatch. A lower score on this test indicates better stair climbing performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, New Taipei City, ROC, Taiwan

IPD SHARING:
Plan to Share IPD: No